CLINICAL TRIAL: NCT03299803
Title: Partnership to Develop and Pilot-Test a Peer Program to Reduce Depressive Symptoms in Men With Physical Disabilities
Brief Title: Depression in Men With Physical Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Dena Hassouneh, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R15NR016362 (NIH)
Record Dates: First submitted 2017-09-25; First posted 2017-10-03 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Men's Healing Pathways (Experimental): Men with physical disabilities will receive a 15 session weekly peer implemented program
  Interventions: Behavioral: Men's Healing Pathways
- Control group (No Intervention): Telephone contact only

INTERVENTIONS:
Behavioral: Men's Healing Pathways — Peer implemented group self management program to reduce depressive symptoms in men with physical disabilities
  Arms: Men's Healing Pathways

SUMMARY:
This project is intended to develop an evidence-based peer group counseling program that addresses depressive symptoms in men with physical disabilities. Expanding treatment options for depressive symptoms in men with physical disabilities will improve their access to care. The benefits of men with physical disabilities receiving effective treatment for depressive symptoms include better health, independent living, and longer life.

DETAILED DESCRIPTION:
Previously the investigators developed, tested and disseminated a highly effective peer counseling program to reduce depressive symptoms in women with physical disabilities (WPDs) in partnership with Oregon Centers for Independent Living (CILs). WPDs with baseline Center for Epidemiologic Depression (CES-D) scores >16 demonstrated significant improvement in depressive symptoms that were sustained over a three month follow-up period (ES partial eta2=.10). The program is offered by two peers in 14 weekly 2.5 hour group sessions. Our academic-disability community partnership created Healing Pathways using community-based participatory research (CBPR) methods and the investigators have sustained our partnership over 9 years. Healing Pathways is currently publicly funded and offered by four of the seven CILs in Oregon. The success of Healing Pathways is a direct result of community investment in and ownership of the program. This project intends to replicate this model to address depression in men with physical disabilities (MPDs).

Depression is a common secondary condition in MPDs, occurring at rates between 37-64%.This is 2-6 times the rate of depression found in non-disabled men. MPDs who work in CILs or other consumer-controlled non-profit agencies are uniquely situated to address depression in their peer group. The Rehabilitation Act of 1973 mandated the formation of CILs to maximize the leadership, empowerment, independence, and productivity of people with disabilities and to integrate them into mainstream society by providing four core independent living services. The core services are: information and referral, independent living skills training, peer counseling, and individual and systems advocacy. CILs are grounded in Independent Living (IL) philosophy, promulgating inclusion across disability-types, de-medicalization and de-institutionalization, and the belief that people with disabilities are the best experts on their own health. There are 403 CILs across the nation, a largely untapped infrastructure with great potential to augment health services for people with disabilities using a peer-to-peer model. The sweeping nature of mental health reforms occurring in the span of a lifetime has given rise to consumer-run peer programs and there is mounting evidence, including randomized controlled trials, that they are efficacious in improving well-being and psychiatric symptoms. Many persons with chronic mental illness prefer peer programs, finding them more relatable and empowering than traditional services. Although many MPDs may also prefer the option of peer counseling compared to traditional psychotherapy, to our knowledge there are no peer programs that address the co-occurrence of physical disability and depression in men. The long-term goal of this program of research is to improve mental health outcomes in people with physical disabilities by partnering with members of this community. This approach recognizes disability communities as cultural entities, respects the values of IL philosophy, and emphasizes the interconnection between mental and physical health. The objective here, the investigators' next step in pursuit of that goal, is to develop and pilot-test a peer program for MPDs with depression. Using a community-engaged, exploratory sequential, mixed methods design, this study intends to achieve the following three specific aims:

1. Adapt the Healing Pathways program to meet the needs of MPDs with depressive symptoms.
2. Conduct a pilot study to assess the feasibility and acceptability of the peer program.
3. Estimate the effect size of the peer program for depressive symptoms. The outcomes of this study will collectively inform the development of a future randomized controlled trial of a program designed to treat depressive symptoms in MPDs. Further, the proposed study addresses several public health goals including Healthy People 2020 goal DH18 to reduce the proportion of people with disabilities who report serious emotional distress,24 and the President's New Freedom Commission on Mental Health goals 1-3, to understand that mental health is essential to overall health, promote mental health treatments that are consumer-driven, and eliminate disparities in mental health care. Because bias against people with disabilities is common among health care providers, education of future health researchers is also necessary to help meet these goals. As part of the proposed project, nursing students will received a mentored experience to support culturally appropriate research with members of the disability community. Experiences will include didactic instruction, community immersion, and research training. Development of a cadre of future researchers who have the knowledge, abilities, and skills to advance the health of people with disabilities through community partnerships is a goal of the project.

ELIGIBILITY:
Inclusion Criteria:

* Self-identifies as having a physical disability
* Diagnosis of Depression
* Must be able to participate and attend all intervention sessions

Exclusion Criteria:

* Currently suicidal with intent and plan
* Diagnosis of schizophrenia or schizoaffective disorder

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 31 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Center for Epidemiologic Studies Depression Measure | 3 months
  20-item self-report measure of depressive symptoms over the past week

CONTACTS AND LOCATIONS:
Locations (1):
- Dena Hassouneh, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No
No information will be shared